CLINICAL TRIAL: NCT01189812
Title: A Randomized, Double-Blind, Placebo-Controlled, Fixed-Dose Study to Assess the Safety and Efficacy of Citalopram in Combination With Lithium or Placebo in the Treatment of Symptoms in Patients With Depressive Mood Disorders
Brief Title: Safety and Efficacy Study of Citalopram and Lithium for the Treatment of Depressive Mood Disorder Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia Northwest Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP-DP-09201
Record Dates: First submitted 2010-03-18; First posted 2010-08-27 (Estimated); Results first posted 2011-06-08 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-08

CONDITIONS: Major Depressive Disorder; Dysthymia; Depression Not Otherwise Specified; Borderline Personality Disorder
Keywords: hopelessness; alone; sad; troubled; depression
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder; Borderline Personality Disorder; Depression | interventions — Lithium Carbonate; Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Citalopram
- Lithium (Active Comparator)
  Interventions: Drug: Lithium Carbonate; Drug: Citalopram

INTERVENTIONS:
Drug: Lithium Carbonate — 300 mg one time per day for 4 weeks
  Arms: Lithium
Drug: Placebo — Take one time daily for 4 weeks
  Arms: sugar pill
Drug: Citalopram — All patients will be administered Citalopram 20 mg to to be taken once daily, by mouth for the duration of the double-blind treatment phase (4 weeks)
  Other Names: Celexa

SUMMARY:
The investigators hypothesize that patients receiving citalopram in combination with lithium will have a greater reduction in depressive symptoms than patients receiving citalopram in combination with placebo.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* Meets criteria for Major Depressive Disorder, Dysthymia, Depression Not Otherwise Specified or Borderline Personality Disorder
* Ability to speak, read and understand the English Language and provide written informed consent

Exclusion Criteria:

* Current, unstable and significant medical condition or illness
* History of Thyroid disorder, seizure disorder, tumors or other CNS condition that predisposes the patient to risk of seizure
* Pregnant or lactating females
* Abnormal clinical laboratory test results
* Intolerance or hypersensitivity to SSRIs or lithium
* History or current diagnosis of bipolar mood disorder, psychosis, schizophrenia or dementia
* Certain mediations my not be used prior or during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arifulla Khan, MD, Principal Investigator — Northwest Clinical Research Center; Vishaal Mehra, MD, Principal Investigator — Aretmis Institute for Clinical Research
Locations (2):
- United States (2):
  - Artemis Institute for Clinical Research, San Diego, California
  - Northwest Clinical Research Center, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 93 patients screened to meet the enrollment target of 80 randomized subjects into this study. Subjects were recruited from two clinical research centers beginning in March 2010. One site was located in Bellevue, WA, and the other in San Diego, CA. The last patient was screened in December 2010.
Pre-assignment Details: After a patients enrolled in the study, the washout period for any excluded concomitant medications was kept to a minimum to avoid potential risk to this severely ill population.
Groups:
- Placebo (Sugar Pill): Patients were administered a 20 mg citalopram tablet in combination with a placebo capsule (sugar pill). Patients were instructed to take medication once daily, by mouth, preferably in the morning.
- Lithium: Patients were administered a 20 mg citalopram tablet in combination with a 300 mg lithium capsule. Patients were instructed to take medication once daily, by mouth, preferably in the morning.
Period: Overall Study
Arm/Group | Placebo (Sugar Pill) | Lithium
Started | 40 | 40
Completed | 32 | 32
Not Completed | 8 | 8
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Out of Window | 4 | 3
Not completed — Moved out of State | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Sugar Pill) | Lithium | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 39 | 78
  >=65 years | 1 | 1 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 38.5 (15.2) | 45.0 (11.6) | 41.8 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 19 | 44
  Male | 15 | 21 | 36
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Sheehan-Suicidality Tracking Scale (S-STS)
Description: The S-STS is an 14 item clinician administered prospective rating scale that scores both treatment-emergent suicidal ideations and suicidal behaviors with scores ranging from 0-40 points. Patients scoring a 0 are experiencing no suicidal thoughts, ideations, or attempts, while a score of 40 indicates a fatal, completed suicide.
  Comparison was made between the citalopram with lithium and the citalopram with placebo treatment groups. Outcome measures are expressed as change scores from the baseline visit to week 4.
Time Frame: 4 weeks; from Baseline to Week 4
Population: The ITT population consisted of 80 patients randomized to lithium (n=40)or placebo (n=40).
Measure: Mean (Standard Deviation); unit: Scores on a Scale (S-STSS)
Units Other Than Participants: Suicidality scales
Arm/Group | Placebo (Sugar Pill) | Lithium
Number analyzed (Participants) | 40 | 40
Number analyzed (Suicidality scales) | 40 | 40
Scores on a Scale (S-STSS) | 4.8 (5.5) | 5.0 (5.1)

2. Secondary Outcome: Beck Hopelessness Scale (BHS)
Description: The BHS measures the extent of negative attitudes about the future. It has particular utility as an indirect indicator of suicidal risk in depressed examinees or individuals who have made suicide attempts.
  Comparison between citalopram and lithium and citalopram and placebo groups in the BHS will be made from baseline to week 4
Time Frame: 4 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Beck Scale for Suicide Ideation (BSS)
Description: The BSS is a 21-item slef-report instrument used to detect ans measure the severity of suicidal ideation in adults. It measures a broad spectrum of attitudes and behaviors for assessing patient suicide risk, as well as reveals specific suicidal characteristics which require greater scrutiny.
  Comparison between citalopram and lithium and citalopram and placebo groups in the BSS will be made from baseline to week 4
Time Frame: 4 weeks
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: Participants

ADVERSE EVENTS:
Time Frame: Adverse event reporting began at the time the patient screened for the study and signed the informed consent document. AEs were collected at each study visit and follow up phone call and could be reported 30 days after last dose of study medication.
Arm/Group | Placebo (Sugar Pill) | Lithium
Serious Adverse Events (participants affected / at risk) | 1/40 | 1/40
Other Adverse Events (participants affected / at risk) | 18/40 | 21/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Sugar Pill) (N=40) | Lithium (N=40)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) — Patient reported that hospitalization post trial participation for worsening depression symptoms.
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Patient was hospitalized for worsening psoriasis during the screening period of the trial.
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Sugar Pill) (N=40) | Lithium (N=40)
Somnolence (Nervous system disorders) | 7 (8) | 6 (6)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (4)
Headaches (Nervous system disorders) | 1 (2) | 9 (11)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Decreased Appetite (Nervous system disorders) | 2 (2) | 2 (2)
Anxiousness (Psychiatric disorders) | 2 (2) | 3 (3)
Restlessness (Nervous system disorders) | 2 (2) | 0 (0)
Common Cold (Infections and infestations) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Upper Respitory Infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No